CLINICAL TRIAL: NCT04656756
Title: Determining the Severity of Physical Symptoms Displayed by Mothers Receiving Personalized Care and Their Level of Perceived Readiness for Discharge After Birth
Brief Title: Determining the Severity of Physical Symptoms Displayed and Their Level of Perceived Readiness for Discharge After Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Durmaz (Other)
Responsible Party: Sponsor-Investigator, Aysegul Durmaz, Asst. Prof., Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Personalized Phy. Symp. Disc.
Record Dates: First submitted 2020-11-29; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Physical Suffering; Post Procedural Discharge
Keywords: Personalized care; Routine care; Postpartum care; Physical symptom; Discharge
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted as a single blind, prospective, and simple randomized controlled trial. The sample was calculated through Power analysis. Consequently, the sample size calculated for α:0.05 and 1-β= 0.95 was 48.Considering the possibility that participants of the sample might be lost or abandon the study, 120 mothers who met the criteria of inclusion to experimental (E) (n=60) and control (C) (n=60) groups were included and assigned to both groups using the permuted block randomization method. The size and number of blocks divided into two groups as E and C was calculated as 20 (3E and 3C) with six mothers in each block. Using Microsoft Office Excel 2013, numbers ranging from 1 to 20 were randomly generated.A total of 120 mothers were evenly and homogeneously assigned to both groups.
Who Masked: Participant
Masking Description: Participants didn't know which group they were allocated. The participants will be blind when they take personalized care from investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The mothers in the experimental group (60) were administered.
  Interventions: Behavioral: Personalized Care
- Control Group (No Intervention): The mothers in the control group (60) were given the routine care.

INTERVENTIONS:
Behavioral: Personalized Care — A clinical and standardized workflow was created for both experimental and control groups. This standardized workflow: consisted of services which included the management of basic medications, routine care regarding the postpartum period, newborn care and health education. After the standardized clinic workflow was formed, a personalized care plan was developed for the experimental group. Each care procedure was shared with the participants in the experimental group. Moreover, all potential alternative care plans were presented to the participants.
  Arms: Experimental Group

SUMMARY:
H1a: There is a difference between the severity of physical symptoms displayed by puerperal women who received routine and personalized care during the early postpartum period.

H1b: There is a difference between the levels of readiness for discharge among puerperal women who received routine and personalized care during the early postpartum period.

H0a: There is no difference between the severity of physical symptoms displayed by puerperal women who received routine and personalized care during the early postpartum period.

H0b: There is no difference between the levels of readiness for discharge among puerperal women who received routine and personalized care during the early postpartum period.

DETAILED DESCRIPTION:
This single-blind randomized controlled trial was conducted between the February and December of 2019. The study was carried out at tertiary care hospital in Turkey. The population of this study consisted of the puerperal women who performed vaginal birth at the maternity unit of a hospital.

Considering the possibility that participants of the sample might be lost or abandon the study, 120 mothers who met the criteria of inclusion to experimental (E) (n=60) and control (C) (n=60) groups were included and assigned to both groups using the permuted block randomization method.The investigators randomly allocated the participants either to the intervention group (which received the personalized care), or to control group (which received the routine care). The mothers in the experimental group (60) were administered personalized care while those in the control group (60) were given the routine care.

The pre-test procedure was performed when the mothers' statuses were stabilized one hour after the admittance to the maternity service. The post-test procedure was conducted one hour before the discharge. Routine care was provided to the mothers in both groups. Routine care means the standard care service provided to mothers following the birth. The standard postpartum basic care components were determined based on the guides and protocols of the hospital. There are three core components of postpartum care regarding the routine care service.

The data were collected using the ''Personal Information Form'', ''Postpartum Physical Symptom Severity Scale'' and ''Perceived Readiness for Discharge After Birth Scale-Form for New Mothers (PRDABS-FNM)''.

Statistical analyses were performed using IBM SPSS (Statistical Package for Social Sciences) Statistics 22 software. Descriptive statistics (mean, standard deviation, frequency and percentage values) were used to assess the results. Kolmogorov-Smirnov test was used to review the goodness of fit to normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* To receive personalized care
* To have vaginal birth
* To have singleton birth
* To be within the early postpartum period (the first 24 hours)
* Not have complications childbirth
* Not have chronic diseases or mental disorders
* Older than 18 years
* To voluntary to participate
* To know how to read, write and speak in Turkish
* To stay within this study until the end
* To fully complete questionnaire
* To have a newborn with no complications
* To have a healthy baby

Exclusion Criteria:

* To receive routine care
* To received theoretical training,
* Not have vaginal birth
* Having multiple birth
* Not to be within the early postpartum period (the first 24 hours)
* Having complications childbirth
* Having chronic diseases or mental disorders
* Younger than 18 years
* To refuse to participate
* Not knowing how to read, write and speak Turkish
* To leave early this study
* Not fill the questionnaire
* Having a newborn with complications
* Having a baby in need of medical care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Pre- Test Severity of Physical Symptoms | 1 hour after the admittance to the maternity service
  Postpartum Physical Symptom Severity Scale; this 4-point Likert scale has 18 items aiming to determine the physical postpartum symptoms. The scale is scored as 0 (none), 1 (mild), 2 (moderate) and 3 (severe). The scale assesses the physical symptoms, such as perineum pain, insomnia, constipation, backpain, headache, hemorrhoid, arthralgia, numbness in hands and feet, vaginal discharge and infection, vaginal bleeding, urinary tract infections, dizziness, varicose vein in legs, urinary incontinence, feeling cold abnormally or coldness in hands and feet, and it evaluates the severity of these symptoms. The total scale score varies between 0 and 54. An increase in the score obtained from the scale indicates high severity of physical postpartum symptoms.
Pre-Test Readiness for Discharge After Birth | 1 hour after the admittance to the maternity service
  Perceived Readiness for Discharge After Birth Scale-Form for New Mothers (PRDABS-FNM); This is a scale assessing the readiness for discharge by mothers' perceptions. It consists of four subdimensions and 23 items. The first item is answered dichotomously (yes/no). The items between 2 and 23 are calculated through the Likert type points ranging from 0 to 10. The subdimensions consisted of 1. Care skills, 2. Expected support; 3. Strength and ability to cope; 4. Stress control and knowledge of accessing help. The lowest and highest scores are 0 and 220. High scores indicate women's readiness for discharge.

SECONDARY OUTCOMES:
Post-Test Severity of Physical Symptoms | 1 hour before the discharge
  Postpartum Physical Symptom Severity Scale; this 4-point Likert scale has 18 items aiming to determine the physical postpartum symptoms. The scale is scored as 0 (none), 1 (mild), 2 (moderate) and 3 (severe). The scale assesses the physical symptoms, such as perineum pain, insomnia, constipation, backpain, headache, hemorrhoid, arthralgia, numbness in hands and feet, vaginal discharge and infection, vaginal bleeding, urinary tract infections, dizziness, varicose vein in legs, urinary incontinence, feeling cold abnormally or coldness in hands and feet, and it evaluates the severity of these symptoms. The total scale score varies between 0 and 54. An increase in the score obtained from the scale indicates high severity of physical postpartum symptoms.
Post-Test Severity of Physical Symptoms | 1 hour before the discharge
  Perceived Readiness for Discharge After Birth Scale-Form for New Mothers (PRDABS-FNM); This is a scale assessing the readiness for discharge by mothers' perceptions. It consists of four subdimensions and 23 items. The first item is answered dichotomously (yes/no). The items between 2 and 23 are calculated through the Likert type points ranging from 0 to 10. The subdimensions consisted of 1. Care skills, 2. Expected support; 3. Strength and ability to cope; 4. Stress control and knowledge of accessing help. The lowest and highest scores are 0 and 220. High scores indicate women's readiness for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Durmaz, Principal Investigator — KSBU
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: If study' IPD are used, my article should be cited.

REFERENCES:
- [Background] Durmaz A, Komurcu N. Relationship Between Maternal Characteristics and Postpartum Hemorrhage: A Meta-Analysis Study. J Nurs Res. 2018 Oct;26(5):362-372. doi: 10.1097/jnr.0000000000000245. PMID 29219937
- [Result] Ceylan B, Eser I. Assessment of individualized nursing care in hospitalized patients in a university hospital in Turkey. J Nurs Manag. 2016 Oct;24(7):954-961. doi: 10.1111/jonm.12400. Epub 2016 Jun 14. PMID 27297976
- [Result] Chien LY, Tai CJ, Hwang FM, Huang CM. Postpartum physical symptoms and depressive symptomatology at 1 month and 1 year after delivery: a longitudinal questionnaire survey. Int J Nurs Stud. 2009 Sep;46(9):1201-8. doi: 10.1016/j.ijnurstu.2009.02.007. Epub 2009 Mar 10. PMID 19278680
- [Result] Finlayson K, Crossland N, Bonet M, Downe S. What matters to women in the postnatal period: A meta-synthesis of qualitative studies. PLoS One. 2020 Apr 22;15(4):e0231415. doi: 10.1371/journal.pone.0231415. eCollection 2020. PMID 32320424
- [Result] Forster DA, McLachlan HL, Davey MA, Biro MA, Farrell T, Gold L, Flood M, Shafiei T, Waldenstrom U. Continuity of care by a primary midwife (caseload midwifery) increases women's satisfaction with antenatal, intrapartum and postpartum care: results from the COSMOS randomised controlled trial. BMC Pregnancy Childbirth. 2016 Feb 3;16:28. doi: 10.1186/s12884-016-0798-y. PMID 26841782
- [Result] Jansson I, Pilhamar E, Forsberg A. Factors and conditions that have an impact in relation to the successful implementation and maintenance of individual care plans. Worldviews Evid Based Nurs. 2011 Jun;8(2):66-75. doi: 10.1111/j.1741-6787.2010.00195.x. Epub 2010 Jun 29. PMID 20604910
- [Result] Johansson M, Thies-Lagergren L, Wells MB. Mothers experiences in relation to a new Swedish postnatal home-based model of midwifery care-A cross-sectional study. Midwifery. 2019 Nov;78:140-149. doi: 10.1016/j.midw.2019.07.010. Epub 2019 Jul 15. PMID 31446229
- [Result] Knier S, Stichler JF, Ferber L, Catterall K. Patients' perceptions of the quality of discharge teaching and readiness for discharge. Rehabil Nurs. 2015 Jan-Feb;40(1):30-9. doi: 10.1002/rnj.164. Epub 2014 Jun 24. PMID 24962625
- [Result] McCarter-Spaulding D, Shea S. Effectiveness of Discharge Education on Postpartum Depression. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):168-72. doi: 10.1097/NMC.0000000000000236. PMID 27128643
- [Result] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Result] Nurhayati N, Songwathana P, Vachprasit R. Surgical patients' experiences of readiness for hospital discharge and perceived quality of discharge teaching in acute care hospitals. J Clin Nurs. 2019 May;28(9-10):1728-1736. doi: 10.1111/jocn.14764. Epub 2019 Feb 6. PMID 30589480
- [Result] Poochikian-Sarkissian S, Sidani S, Ferguson-Pare M, Doran D. Examining the relationship between patient-centred care and outcomes. Can J Neurosci Nurs. 2010;32(4):14-21. PMID 21268489